CLINICAL TRIAL: NCT01185886
Title: Translational Research - Observational Study for Identification of New Possible Prognostic Factors and Future Therapeutic Targets in Children With Acute Lymphoblastic Leukemia (ALL)
Brief Title: Study of Blood and Tissue Samples in Children With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-58081; EORTC-58081; EU-21057
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Leukemia; Lymphoma
Keywords: untreated childhood acute lymphoblastic leukemia; L1 childhood acute lymphoblastic leukemia; L2 childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; Philadelphia chromosome positive childhood precursor acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Gene Expression Profiling; Amplified Fragment Length Polymorphism Analysis; Pharmacogenomic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: mutation analysis
Genetic: polymorphism analysis
Other: biologic sample preservation procedure
Other: laboratory biomarker analysis
Other: pharmacogenomic studies

SUMMARY:
RATIONALE: Collecting and storing samples of tumor tissue, blood, bone marrow, and other body fluids from patients to test in the laboratory and collecting information about the patient's health and treatment may help doctors learn more about cancer and help the study of cancer in the future. Studying these samples in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment.

PURPOSE: This research study is collecting and looking at blood and tissue samples in children with newly diagnosed acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Collect clinical data in parallel with biological data and samples from children with newly diagnosed acute lymphoblastic leukemia for biobanking, and use part of the biobanked material to perform specific translational projects to achieve objectives II-IV.
* To identify new prognostic factors (e.g., minimal-residual disease [MRD] significance in small subgroups, miRNAs expression profile, PAX5 mutation, genetic abnormalities in T-cell acute lymphoblastic leukemia [T-ALL], and RAS pathway activation) and future therapeutic targets in children with newly diagnosed acute lymphoblastic leukemia.
* To identify leukemia cell genetic alterations (e.g., mutations in T-ALL and miRNA expression in B-cell acute lymphoblastic leukemia [B-ALL]) and related molecular pathways (e.g., RAS pathway) underlying leukemogenesis.
* To identify patient pharmacogenetic polymorphisms impacting individual response to corticosteroids as part of standard therapy and investigate their prognostic significance.

OUTLINE: This is a prospective observational biobanking study.

Patients undergo clinical evaluation, laboratory tests, and imaging periodically. Data are collected before, during, and after first-line standard therapy. Clinical data are collected from all patients in parallel with the biological data and samples. Biological samples are partly used to perform specific translational research (TR) projects. Remaining biological materials are stored for future research.

The following TR projects are performed on the biological samples for this study. Biological samples are analyzed for allele-specific amplification of Ig/TCR clonal rearrangements to quantify minimal-residual disease (MRD) via real-time PCR (TR1 Project); miRNA expression via qPCR (TR 2 Project); the detection of main point mutations via high-resolution melting PCR (TR 3 Project); genetic polymorphisms via real-time TaqMan allelic-discrimination method (TR 4 Project); clinical significance of genetic abnormalities via quantitative real-time RT-PCR, direct sequencing, and fluorescence in situ hybridization (TR 5 Project); and RAS pathway activation via single-nucleotide polymorphism (SNP) analysis and gene-expression analysis (TR 6 Project).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute lymphoblastic leukemia (ALL), meeting the following criteria:

  * FAB L1 or L2 morphology (any immunophenotype) and acute leukemias of ambiguous lineage (including biphenotypic or bilineal acute lymphoblastic leukemia)

    * Patients with mature B-cell acute lymphoblastic leukemia (B-ALL) (FAB L3 morphology and immunophenotypical mature B phenotype or B-ALL with documented presence of karyotype t(8;14), t(2;8) t(8;22) or breakpoints as in mature B-ALL) are excluded from this study
* Patients must also meet the following criteria for participating in individual translational research (TR) project:

  * TR 1 project (MRD prognostic significance in small ALL subgroups):

    * All patients, categorized according to response to pre-phase (< or > 1,000 peripheral blasts/mm³ at day 8) and minimal-residual disease (MRD) level at end of the induction therapy
    * iAmp(21q) detected at presentation
    * Hypodiploidy detected at presentation by karyotype and/or fluorescence in situ hybridization (FISH) and/or DNA index
  * TR 2 project (miRNAs expression in pediatric ALL):

    * Initially, average-risk 1 (AR1) patients
    * In a second stage, the analysis might be extended to low-risk patients that still show treatment failure and high-risk ALL patients
  * TR 3 project (Prognostic value of newly described mutations in childhood B-ALL)

    * Initially, only B-cell precursor ALL patients
  * TR 4 project (Pharmacogenetics of the response to prephase and induction therapy):

    * All ALL patients
  * TR 5 project (Clinical significance of genetic abnormalities in childhood T-ALL) :

    * All patients with T-cell ALL, as defined by expression of T-cell surface antigens
  * TR 6 project (RAS pathway activation in childhood B-ALL):

    * All patients with B-lineage ALL
* Patients with Philadelphia-chromosome positive ALL (documented presence of t(9;22)(q34;q11) and/or of the BCR/ABL fusion transcript) are eligible
* Scheduled to receive therapy as per institutional standard practice and have not started therapy (except for a maximum of 7 days of systemic corticosteroids prior to diagnosis)
* May only be registered to this study once

PATIENT CHARACTERISTICS:

* No psychological, familial, sociological, or geographical condition potentially hampering participation in the study protocol and follow-up schedule
* Patients with Down syndrome are eligible

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival
Disease-free interval from complete remission
Response to pre-phase standard therapy
Adverse events to induction standard therapy
Overall survival
Biomarker levels

CONTACTS AND LOCATIONS:
Overall Officials: Helene Cave, Principal Investigator — CHU - Hopital Robert Debre; Yves Benoit, MD, Principal Investigator — University Ghent; Yves Bertrand, MD, Principal Investigator — Hospices Civils de Lyon
Locations (21):
- Belgium (7):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hopital Universitaire Des Enfants Reine Fabiola, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Regional De La Citadelle, Liège
- France (13):
  - CHRU de Besancon - Hopital Saint-Jacques, Besançon
  - CHU de Caen - Hopital Cote de Nacre, Caen
  - CHU de Grenoble - La Tronche - Hôpital A. Michallon, Grenoble
  - CHRU de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Hopital Arnaud De Villeneuve, Montpellier
  - CHU de Nice - Hopital De L'Archet, Nice
  - CHU - Hopital Robert Debre, Paris
  - Hopital Jean Bernard, Poitiers
  - CHU de Reims - American Memorial Hospital, Reims
  - Centre Hospitalier Félix Guyon, Saint-Denis
  - Hopitaux Universitaires de Strasbourg - Hautepierre, Strasbourg
  - CHU de Toulouse - C.H.U. De Toulouse - Hopital Des Enfants, Toulouse
- Instituto Portugues De Oncologia - Centro Do Porto, Porto, Portugal

REFERENCES:
- [Derived] Matthijssens F, Sharma ND, Nysus M, Nickl CK, Kang H, Perez DR, Lintermans B, Van Loocke W, Roels J, Peirs S, Demoen L, Pieters T, Reunes L, Lammens T, De Moerloose B, Van Nieuwerburgh F, Deforce DL, Cheung LC, Kotecha RS, Risseeuw MD, Van Calenbergh S, Takarada T, Yoneda Y, van Delft FW, Lock RB, Merkley SD, Chigaev A, Sklar LA, Mullighan CG, Loh ML, Winter SS, Hunger SP, Goossens S, Castillo EF, Ornatowski W, Van Vlierberghe P, Matlawska-Wasowska K. RUNX2 regulates leukemic cell metabolism and chemotaxis in high-risk T cell acute lymphoblastic leukemia. J Clin Invest. 2021 Mar 15;131(6):e141566. doi: 10.1172/JCI141566. PMID 33555272